CLINICAL TRIAL: NCT07292480
Title: Monthly Monitoring of Plasma NfL in Treated RRMS to Detect Persistent Infraclinical Disease Activity
Brief Title: Monthly Monitoring of Plasma NfL in Treated Relapsing-remitting Multiple Sclerosis to Detect Persistent Infraclinical Disease Activity
Acronym: MoMo-NfL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FINEX/2025/ET-01
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting
Keywords: Biomarker
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pNfL monitoring group (Experimental)
  Interventions: Other: Monthly pNfL monitoring
- Standard care (No Intervention)

INTERVENTIONS:
Other: Monthly pNfL monitoring — Monthly pNfL monitoring from blood samples. In case of >50% pNfL increase as compared to the mean of the 2 previous measures, an unscheduled visit with brain and spinal cord MRI will be scheduled
  Arms: pNfL monitoring group

SUMMARY:
Reference MRI scan is recommended 6 months after treatment onset in patients with multiple sclerosis (MS), and follow-up scans at 12 months later to monitor subclinical activity. When monitoring treatment response in patients treated with disease modifying treatments (DMTs), the measurement of new or enlarging T2/FLAIR hyperintense lesions (NELs) is the preferred MRI method supplemented by contrast-enhancing lesions (CELs) for monitoring treatment response. However, some studies have suggested the deposition of gadolinium-based contrast agents in the basal ganglia and dentate nucleus of patients who underwent serial MRI acquisitions. Although significant clinical consequences of these deposits have not been demonstrated, further studies are required to better understand the potential long-term biological and clinical effects of gadolinium administration. To circumvent this potential risk, several recommendations suggested avoiding unnecessary use of gadolinium for follow-up scans. New sequences are also developed to replace gadolinium injection for the detection of active lesions. Moreover, MRI remains costly and time-consuming. In addition, systematic yearly MRI monitoring is not adapted to detect silent active lesions. This can delay identification of treatment failure and increase the risk of relapses and disability worsening, especially in the context of escalation therapy.

Therefore, biological markers could allow more frequent analysis of disease activity and detect treatment failure earlier than classical clinical and MRI monitoring. Their use would greatly help clinicians to switch for high efficacy treatments (HET) and avoid potential relapses.

Measurement of a structural axonal protein, neurofilament, in serum or plasma has shown promise as a marker of neuroaxonal injury and a measure of treatment response. In MS, cerebrospinal fluid (CSF) neurofilament-light chain (NfL) is also increased and is positively associated with MRI lesion load and disability scores and is a marker of treatment response.

WThe study authors hypothesize that monthly plasma neurofilament-light chain (pNfL) monitoring can sensitively highlight subclinical (radiological disease activity) RDA by performing early MRI scans to confirm EDA and lead to timely treatment escalation.

The main objective of this study is to compare the time to EDA in both arms (monthly pNfL monitoring vs. standard care with regular MRI scans), in patients with EDA.

ELIGIBILITY:
Inclusion Criteria:

* Patient with RRMS according to 2017 McDonald's criteria.
* Less than 5 years from disease onset.
* Active RRMS (EDA) observed during the last 24 months: relapse and/or NELs and/or CELs as compared to a previous MRI performed within 24 months (± 3 months).
* MET (IFN, GA, TE, fumarates) for less than 24 months.
* Standard MRI follow-up scan performed less than 30 days before inclusion.
* Clinically stable disease for at least 30 days.
* Patients included in observational studies and cohorts (OFSEP, PROMISE …) will be eligible for inclusion in MoMo-NfL.
* For women with reproductive potential: negative pregnancy test at the time of inclusion and use of an effective method to avoid pregnancy for the duration of the trial.
* Patients able to adhere to the study visit schedule.
* Patient must have signed and given the consent.
* Patient affiliated or beneficiary of a health insurance plan.

Exclusion Criteria:

* Pregnant or breastfeeding woman.
* Patient unable to perform brain and/or spinal cord MRI scans.
* Patient not willing to perform monthly blood punctures.
* Patient treated with HET (S1P agonists, natalizumab, ocrelizumab, ofatumumab, rituximab, alemtuzumab, cladribine, mitoxantrone).
* Patient with a relapse within 6 months before inclusion.
* Patient with CELs within 3 months before inclusion.
* Patient with progressive MS.
* Patient unable to sign the consent.
* It is impossible to correctly inform the patient.
* Patient being involved or having been involved in an interventional research (RIPH type 1 or drug research or clinical investigation of medical device) 3 months before the inclusion visit.
* Patient under judicial protection, or is an adult under guardianship.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control for the duration of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Time to evidence of disease activity between groups | Month 12
  As assessed by new relapse and/or occurrence of NELs and/or CELs on a follow-up MRI scan
Time to evidence of disease activity between groups | Month 24
  As assessed by new relapse and/or occurrence of NELs and/or CELs on a follow-up MRI scan

SECONDARY OUTCOMES:
Proportion of CELs between groups | Month 12
  percent of active (contrast-enhancing) lesion
Proportion of CELs between groups | Month 24
  percent of active (contrast-enhancing) lesion
Rate of clinical relapses between groups | Month 12
  percentage patients experiencing relapse
Rate of clinical relapses between groups | Month 24
  percentage patients experiencing relapse
Time to switch to high efficacy treatments | Month 12
  Days
Time to switch to high efficacy treatments | Month 24
  Days
Proportion of patients switching to high efficacy treatments between groups | Month 12
  Percentage
Proportion of patients switching to high efficacy treatments between groups | Month 24
  Percentage
Change in pNfL levels in patients experiencing relapse with active MRI in experimental group | Upon experiencing relapse (maximum Month 24)
  pg/mL; measured using Lumipulse® G NfL Blood
Change in pNfL levels in patients experiencing acute clinical event in experimental group | Upon experiencing an acute clinical event (maximum Month 24)
  pg/mL; measured using Lumipulse® G NfL Blood
Change in pNfL levels in patients experiencing radiological disease activity without clinical symptoms in experimental group | Upon experiencing radiological disease activity (maximum Month 24)
  pg/mL; measured using Lumipulse® G NfL Blood
Change in pNfL levels in patients switching to high efficacy treatments | Upon evidence of disease activity (maximum Month 24)
  pg/mL; measured using Lumipulse® G NfL Blood

OTHER OUTCOMES:
To estimate the best threshold of pNfL increase (last measure as compared to the mean of 2 previous measures) with best accuracy to detect evidence of disease activity | Month 24
  pNfL levels in pg/mL
Time to evidence of disease activity using optimized threshold in experimental group | Month 24
  Months
Correlation between basal pNfL fluctuations in patients with no evidence of disease activity and brain health questionnaire score | Month 24
  Brain-Q
Description of adverse events | Month 24
  Descriptive
Level of disability | Baseline (Day 0)
  EDSS (Extanded Disability Status Scale) score, range: 0.0-10
Level of disability | Month 12
  EDSS (Extanded Disability Status Scale) score, range: 0.0-10
Level of disability | Month 24
  EDSS (Extanded Disability Status Scale) score, range: 0.0-10
Information processing speed impairment | Baseline (Day 0)
  CSCT (Computerized Speed Cognitive Test): score and standard deviation
Information processing speed impairment | Month 12
  CSCT (Computerized Speed Cognitive Test): score and standard deviation
Information processing speed impairment | Month 24
  CSCT (Computerized Speed Cognitive Test): score and standard deviation
Manual dexterity | Baseline (Day 0)
  NHPT (Nine Hole Peg Test): time (seconds)
Manual dexterity | Month 12
  NHPT (Nine Hole Peg Test): time (seconds)
Manual dexterity | Month 24
  NHPT (Nine Hole Peg Test): time (seconds)
Walking function | Baseline (Day 0)
  T25FW (Timed 25-Foot Walk); time (seconds)
Walking function | Month 12
  T25FW (Timed 25-Foot Walk); time (seconds)
Walking function | Month 24
  T25FW (Timed 25-Foot Walk); time (seconds)
Patient-reported change in status | Baseline (Day 0)
  PGIC (Patient Global Impression of Change scale): score (7 points Likert scale)
Patient-reported change in status | Month 12
  PGIC (Patient Global Impression of Change scale): score (7 points Likert scale)
Patient-reported change in status | Month 24
  PGIC (Patient Global Impression of Change scale): score (7 points Likert scale)
Patient-reported quality of life | Baseline (Day 0)
  EQ-5D-5L score (0-100)
Patient-reported quality of life | Month 12
  EQ-5D-5L score (0-100)
Patient-reported quality of life | Month 24
  EQ-5D-5L score (0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvenot, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France